CLINICAL TRIAL: NCT05006079
Title: Opioid/Benzodiazepine Polydrug Abuse: Integrating Research on Mechanisms, Treatment and Policies - Study 3
Brief Title: Opioid/Benzodiazepine Polydrug Abuse: Aim 3
Acronym: MAP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Mark Greenwald, PhD, Professor of Psychiatry and Behavioral Neurosciences; and Director, Substance Abuse Research Division, Wayne State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB-21-07-3844
Record Dates: First submitted 2021-08-04; First posted 2021-08-16 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Opioid Abuse; Benzodiazepine Abuse; Polysubstance Abuse
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Morphine; Alprazolam

STUDY DESIGN:
Intervention Model Description: Repeated measures, placebo-controlled, randomized crossover
Who Masked: Participant, Outcomes Assessor
Masking Description: drug doses will be encapsulated, and placebo is included in the design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Placebo drug (Placebo Comparator): Lactose, administered both at 9:30 am and 12:00 pm
  Interventions: Drug: Placebo
- Morphine alone (Active Comparator): 15mg immediate-release oral morphine, administered both at 9:30 am and 12:00 pm
  Interventions: Drug: Morphine
- Alprazolam alone (Active Comparator): 0.25mg oral alprazolam, administered at both 9:30 am and 12:00 pm
  Interventions: Drug: Alprazolam
- Morphine then alprazolam (Active Comparator): 15mg oral morphine administered at 9:30 am, then 0.25mg oral alprazolam administered at 12:00 pm
  Interventions: Drug: Morphine; Drug: Alprazolam
- Alprazolam then morphine (Active Comparator): 0.25mg oral alprazolam administered at 9:30 am, then 15mg oral morphine administered at 12:00 pm
  Interventions: Drug: Morphine; Drug: Alprazolam
- Morphine+alprazolam simultaneously (Active Comparator): morphine 15mg + 0.25mg alprazolam at 9:30 am, then morphine 15mg + 0.25mg alprazolam at 12:00 pm
  Interventions: Drug: Morphine; Drug: Alprazolam

INTERVENTIONS:
Drug: Morphine — immediate release oral 15mg dose
  Arms: Alprazolam then morphine; Morphine alone; Morphine then alprazolam; Morphine+alprazolam simultaneously
Drug: Alprazolam — oral 0.25mg dose
  Arms: Alprazolam alone; Alprazolam then morphine; Morphine then alprazolam; Morphine+alprazolam simultaneously
Drug: Placebo — Lactose
  Arms: Placebo drug

SUMMARY:
In this study, the investigators will measure affective, neurocognitive and behavioral outcomes related to chronic use of opioids and benzodiazepines (screening phase), and in response to the administration of the opioid morphine, the benzodiazepine alprazolam, morphine then alprazolam, alprazolam then morphine, morphine+alprazolam simultaneously, and placebo (laboratory pharmacology experiment). The latter will enable the investigators to assess the effects of an opioid alone, benzodiazepine alone, concurrent and simultaneous administration of opioid+benzodiazepine, relative to a placebo control.

DETAILED DESCRIPTION:
The investigators propose that benzodiazepine/opioid polysubstance abuse is perpetuated by a dual-deficit in affective/hedonic regulation (difficulties modulating emotional reactions relative to the context and the person's long-term goals). Furthermore, the investigators propose that this dual-deficit biases neurocognition (interferes with executive function) and behaviors (guided by negative reinforcement processes such that polysubstance use acutely blunts aversive states and directs actions away from natural rewards). The scientific premise for this project builds on George Koob's foundational concept that addiction is a 'reward-deficit/stress-surfeit disorder'. There is an urgent need to obtain clinical pharmacology and mechanistic data to test this hypothesis of dual-deficit in affective/hedonic regulation. This study will use human laboratory methods to test affective, neurocognitive and behavioral mechanisms that maintain benzodiazepine/opioid polysubstance abuse.

The screening phase of this human laboratory study will include measures of affective dysregulation related to benzodiazepine/opioid polysubstance use behaviors. These include distress tolerance, pain sensitivity and nocebo responding, and biomarkers (e.g. plasma cortisol). Also, the investigators will include behavioral measures of drug and non-drug reinforcement (e.g. economic simulations of price elasticity of alprazolam and morphine) and neurocognition (e.g. drug attentional bias, response inhibition, cognitive flexibility).

During the pharmacology study the investigators will administer oral placebo, morphine alone and alprazolam doses alone, as well as morphine and alprazolam sequentially (in counterbalanced order) and simultaneously. Following each drug administration, the investigators will measure responses in affective (e.g. anxiety levels, distress tolerance), neurocognitive (e.g. executive function, learning) and behavioral domains (e.g. impulsivity, psychomotor function, reinforcer preferences). The lab study is highly significant because we lack prospective, controlled, dose-response studies that identify whether opioids, benzodiazepines, and their combination modulate core phenotypes that underlie this harmful polysubstance abuse. Testing effects of both sequential and simultaneous benzodiazepine/opioid administration within the same individuals will establish a firm foundation for understanding which phenotypes are sensitive to disruption and may respond to treatment.

Findings from this study will help to focus clinical assessment and identify mechanisms that maintain benzodiazepine/opioid polysubstance abuse, toward the development of novel medication-assisted, evidence-based psychosocial interventions.

ELIGIBILITY:
Inclusion Criteria:

* must self-report past 10-year experience taking opioid and sedative drugs (for therapeutic or non-therapeutic reasons), but not necessarily at the same time. As an alternative to the sedative drug exposure requirement, participants must have used alcohol on at least 3 separate days during the past month. Participants may have current mild- or moderate-severity Opioid Use Disorder or current mild- or moderate-severity Sedative Use Disorder;
* must not be seeking treatment for their substance use problems;
* must be in current good overall health

Exclusion Criteria:

* meet DSM-5 criteria for current psychosis, bipolar disorder, or severe depression (i.e. severe psychiatric disorder);
* meet DSM-5 criteria for severe substance use disorder for any substance (e.g. Sedative, Opioid, Alcohol);
* past-month benzodiazepine or opioid prescription (which would suggest daily use, tolerance, or withdrawal upon cessation);
* report of past-year any-drug overdose or suicide attempt/ideation;
* exhibit cognitive impairment (IQ < 80 on the Shipley Institute of Living Scale);
* neurological, cardiovascular, pulmonary, or systemic diseases (see specific exclusionary conditions under Protection of Human Subjects);
* body mass index > 38 kg/m2;
* females who are pregnant (urine), lactating or heterosexually active (self-report) and not using medically approved birth control;
* treatment with methadone, buprenorphine or naltrexone;
* past 30-day use of contraindicated medications;
* alcohol-positive breath sample (>.02% breath alcohol concentration);
* urine sample positive for methadone, cocaine, amphetamines, or barbiturates (<300 ng/ml)
* intolerance of lactose

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
State anxiety | within-session peak change from pre-drug baseline to 15-120 min post-drug 1 and 15-240 min post-drug 2 administration; measured in each of the 6 laboratory sessions over about 3 weeks
  State Trait Anxiety Inventory - state anxiety scale total score
Positive affect | within-session peak change from baseline to 15-120 min post-drug 1 and 15-240 min post-drug 2 administration; measured in each of the 6 laboratory sessions over about 3 weeks
  Positive and Negative Affect Scale-Short Form (PANAS-SF) positive affect scale score
Negative affect | within-session peak change from baseline to 15-120 min post-drug 1 and 15-240 min post-drug 2 administration; measured in each of the 6 laboratory sessions over about 3 weeks
  Positive and Negative Affect Scale-Short Form (PANAS-SF) negative affect scale score

SECONDARY OUTCOMES:
Symbol matching performance task | difference from placebo condition, measured within each session at 15-240 min post-drug 2 administration; measured in each of the 6 laboratory sessions over about 3 weeks
  Digit Symbol Substitution Task (DSST) symbol matching total score
Impulsivity performance task accuracy | difference from placebo condition, measured within each session at 15-240 min post-drug 2 administration; measured in each of the 6 laboratory sessions over about 3 weeks
  Go/No task percentage of trials correct
Cognitive flexibility performance task | difference from placebo condition, measured within each session at 15-240 min post-drug 2 administration; measured in each of the 6 laboratory sessions over about 3 weeks
  Wisconsin Card Sorting Task (WCST) percentage of trials correct
Cognitive inhibition performance task | difference from placebo condition, measured within each session at 15-240 min post-drug 2 administration; measured in each of the 6 laboratory sessions over about 3 weeks
  Addiction Stroop Task, reaction time to drug vs. neutral words presented in different colors
Vigilance performance task | difference from placebo condition, measured within each session at 15-240 min post-drug 2 administration; measured in each of the 6 laboratory sessions over about 3 weeks
  Psychomotor Vigilance Task (PVT) average reaction time
Hypothetical drug purchasing questionnaire | difference from placebo condition, measured within each session at 15-240 min post-drug 2 administration; measured in each of the 6 laboratory sessions over about 3 weeks
  Intensity and elasticity of drug demand. This is measured by having the participant make a series of independent choices as to how many drug units s/he will purchase across a range of (low to high) unit prices. Demand intensity is the drug purchase amount at the lowest non-zero price. Demand intensity is the calculated point on the price/purchasing curve where the slope (in log/log space) equals -1 (i.e. 'tipping point' where purchasing decreases more rapidly than the rate of increase in drug price).
Preference for natural reinforcement choice procedure | difference from placebo condition, measured within each session at 15-240 min post-drug 2 administration; measured in each of the 6 laboratory sessions over about 3 weeks
  Number of choices for money vs. avoiding listening to soundtrack of crying babies
Monetary delay discounting questionnaire | difference from placebo condition, measured within each session at 15-240 min post-drug 2 administration; measured in each of the 6 laboratory sessions over about 3 weeks
  Participants are asked to make a series of independent choices (preferences) for delayed larger amounts of money vs. smaller immediate amounts of money. The outcome is the rate at which future choice value is discounted, measured by area under the time-delay curve
Respiration rate | within-session peak change from baseline to 15-120 min post-drug 1 and 15-240 min post-drug 2 administration; measured in each of the 6 laboratory sessions over about 3 weeks
  Breaths per minute, measured by behavioral observation
Oxygen saturation | within-session peak change from baseline to 15-120 min post-drug 1 and 15-240 min post-drug 2 administration; measured in each of the 6 laboratory sessions over about 3 weeks
  Percentage oxygen saturation, measured by photoplethysmograph
Heart rate | within-session peak change from baseline to 15-120 min post-drug 1 and 15-240 min post-drug 2 administration; measured in each of the 6 laboratory sessions over about 3 weeks
  Pulse rate (beats per minute), measured by photoplethysmograph
Blood pressure | within-session peak change from baseline to 15-120 min post-drug 1 and 15-240 min post-drug 2 administration; measured in each of the 6 laboratory sessions over about 3 weeks
  Systolic and diastolic blood pressure (mm Hg)
Pupil diameter | within-session peak change from baseline to 15-120 min post-drug 1 and 15-240 min post-drug 2 administration; measured in each of the 6 laboratory sessions over about 3 weeks
  Pupil size (mm), measured by digital photography
Drug effect visual analog scale (VAS) ratings | within-session peak change from baseline to 15-120 min post-drug 1 and 15-240 min post-drug 2 administration; measured in each of the 6 laboratory sessions over about 3 weeks
  0-100 scale ratings of alert, difficulty concentrating, clumsy, confused, forgetful, blurred vision, dizzy, heaviness in limbs, mellow, yawning, stimulated, sedated, sleepy, tired, energetic, self-confident, dreamy, floating, sluggish, tingling, high, liking, good drug effect, bad drug effect
Drug craving visual analog scale (VAS) ratings | within-session peak change from baseline to 15-120 min post-drug 1 and 15-240 min post-drug 2 administration; measured in each of the 6 laboratory sessions over about 3 weeks
  0-100 scale rating of "want to take drug again", "desire to use", and "craving" for opioids, sedatives, alcohol, cigarettes, marihuana, and cocaine
Sleep efficiency | difference from placebo condition, measured on an outpatient basis during the evening after each laboratory drug administration; measured after each of the 6 laboratory sessions over about 3 weeks
  Percentage of sleep time (time asleep divided by time in bed), measured using WatchPat device

CONTACTS AND LOCATIONS:
Overall Officials: Mark K Greenwald, PhD, Principal Investigator — Wayne State University
Locations (1):
- Tolan Park Medical Building, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.